CLINICAL TRIAL: NCT03555058
Title: Comprehensive individUalized pRoactive ThErapy of Crohn's Disease Trial: The CURE-CD Trial
Brief Title: The CURE - CD Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Shomron BenHorin, Prof., Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4945-18-SMC
Record Dates: First submitted 2018-05-27; First posted 2018-06-13 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: CD - Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High risk- TDM (Other): Treatment escalation per TDM and physician's decision.
  Interventions: Other: Treatment escalation
- High risk- Follow Up (No Intervention): Patients randomized to this arm will keep with the follow-up regime. Treatment escalation will occur only upon worsening of symptoms.
- Low risk (No Intervention): Control group. Patients will be assigned to this group based on VCE results and will not undergo randomization.

INTERVENTIONS:
Other: Treatment escalation — Treatment escalation per TDM and physician's decision.
  Arms: High risk- TDM

SUMMARY:
A prospective randomized three-arms controlled trial of Crohn's Disease (CD) patients in remission of <24 months duration. Patients will undergo screening by Magnetic Resonance Enterography (MRE) and patency capsule, and (if agreeing by separate consent) a baseline colonoscopy. Patients in whom patency of small bowel is proven will undergo video-capsule using the dedicated Inflammatory-Bowel Disease (IBD)-capsule (PillCam Crohn's). Patients with Lewis score>350 for worst small bowel segment will be classified as high-risk and will be randomized for continued standard treatment or proactive treatment. Proactive treatment will consist of escalating/switching biologic treatment according to the pre-defined therapeutic drug monitoring (TDM)-based treatment-intensification protocol, or will consist of initiating biologic therapy in high-risk patients not receiving biologics at the time of enrollment. Both high-risk patients arms - the continued standard treatment and the proactive arm - will be followed up by clinic visits with physical examination, inflammatory and immune markers' assessment and microbiome analysis every 3 months and by serial video-capsule endoscopy (VCE) studies+ intestinal UltraSound (US) every six months. Patients who are classified as low-risk patients, as per Lewis score<350 at baseline, will continue standard treatment and be similarly followed. All enrolled patients will undergo MRE at the end of the trial. All patients will undergo in addition blood and stool sampling for inflammatory markers, immune-phenotyping and microbiome analysis. All patients will undergo MRE at the end of the trial.

DETAILED DESCRIPTION:
1. Entry procedures: Patients will undergo clinical examination and history taking and then will undergo patency capsule. If patency is proven, patients will undergo a third generation pan-enteric capsule endoscopy (PillCam Crohn), ileocolonoscopy with biopsies (by separate consent), MRE, Intestinal US, biomarkers, immune & microbiome analysis, and health related quality of life assessment and patient reported outcome (PRO) standard questionnaires. (see Appendix 1 for complete protocol of baseline pan-enteric capsule endoscopy and ileocolonoscopy evaluation, Appendix 2 for complete protocol of MRE examination, Appendix 3 for blood and stool sample collection protocols, Appendix 4 for Intestinal US protocol, appendix 5 for microbiomic analysis protocol, appendix 6 for health related quality of life/cost assessments, appendix 7 for Immune analysis).
2. Follow-up procedures: Capsule endoscopy, nutritional and intestinal US studies will be performed every 6 months for the total study duration of 2 years. For patients with only small bowel disease these will be without preparation. Additionally, periodic (every 3 months) assessment will be performed for inflammatory, microbiome, imaging attributes, quality of life and immunophenotyping, as outlined below in description of tasks for work packages.
3. Risk stratification and outcomes: Based on VCE results and according to the predictive algorithm defined by the first project's results, patients will be classified as high risk if having Lewis score (LS) ≥350 for the small bowel tertile with the highest score, or as having low risk (LS<350 highest tertile score) for future relapse of disease.

Low risk patients will continue the monitoring scheme and their treatment regimen unaltered. Patients with LS ≥350 will be randomized to either continue follow-up with unaltered therapy or to proactive therapy optimization with TDM assessment. Therapy will be optimized based on the optimization protocol described below, with the aim to prevent flares and complications. Follow up to determine the occurrence of clinical flares and complications as well as the status of inflammatory process will be performed for all patients q3months. Study will be terminated and a patient will be withdrawn upon disease flare or complication or if a change of CD medications was instituted (except for treating verified infectious complication such as C. difficile infection) and such a patient will be considered a non-responder. A patient will also be withdrawn if in the opinion of the Principle Investigator (PI), a new adverse event or medical condition is present that endangers the patient's wellbeing if the study protocol is adhered to. To maintain temporally-restricted blinding, VCE results will be disclosed up to three months following the performance of VCE.

* In a sub-group of consenting patients, stool samples for microbiome analysis (see below) will be collected daily for a designated period of time. In a sub-group of consenting patients, additional on-line data collection methods will be employed (see below).

Risk-based intervention: Patients meeting the VCE-based high-risk criteria and who were randomized to proactive treatment arm will receive therapy intensification within 30 days. Re-assessment of response to the intensified therapy will be performed by repeated VCE and bio-markers after 6 months. The intensification protocol will be as appears below. Briefly, patients receiving immunomodulators,5-Aminosalicylates (5ASA) or no treatment at the time they are found to have high risk of imminent flare or complication will receive induction with a biologic of the anti-Tumor necrosis Factor (TNF)- Infliximab (IFX), Adalimumab (ADA)- or anti-integrin (VDZ) classes as per standard induction protocols for these agents. The choice of the biologic will be guided by the treating physician's discretion as per the individual patient-related considerations. In patients already on a biologic, intervention will be guided by protocolized TDM results for patients on anti-TNFs, whereas patients receiving vedolizumab will first receive an interval-halving intervention. Protocolized anti-TNF TDM-based intervention will comprise of increasing the dose of anti-TNF, or switching anti-TNF, or switching out-of-class according to the drug/anti-drug antibodies thresholds and algorithms set by previous works by our group in this field, using the same assay that will be employed in the present trial. Re-adjustment of therapy according to these principles will be performed if 6-month VCE re-assessment does not show a reduction of patient risk score to the range of a low risk VCE-based score. Patients who received an intervention and in whom follow-up 6 months VCE does not show a reduction of 225 points on the Lewis score or highest segment Lewis score of <350, will receive the next protocolized drug optimization.

Intervention protocol in proactive arm based on current treatment and TDM finding:

ADL with drug level<8mcg/ml/AAA<4mcg/ml-eq ADL dose-doubling ADL with drug level <8mcg/ml/AAA>4mcg/ml-eq Switch anti TNF or add IMM ADL with drug level >8mcg/ml Switch out of class IFX with drug level <6mcg/ml/ATI<9mcg/ml-eq IFX dose-doubling IFX with drug level <6mcg/ml/ATI>9mcg/ml-eq Switch anti TNF or add IMM IFX with drug level >6mcg/ml Switch out of class VDZ e/8 week VDZ interval halving VDZ e4W/CD3CD45RO target occupied >85% Switch out of class VDZ e4W/ CD3CD45RO target occupied<85% VDZ double-dosing 600/4w UST 90mg/SC e12w or e/8W Shorten interval e/4w No treatment, 5-ASA or AZA/6MP >> Start biologic ADL - adalimumab, IFX- infliximab, VDZ - vedolizumab UST - Ustekinumab AAA- antibodies to adalimumab, ATI antibodies to infliximab, IMM - immunomodulator

ELIGIBILITY:
Inclusion Criteria:

* CD patients in steroid-free remission for at least 3 months, but no more than 2 years.
* CDAI < 150.

Exclusion Criteria:

* Clinical remission for more than 2 years.
* Patients on a second/third line of biologic class of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Rate of disease flares/complications in high-risk patients | 24 months
  The rate of disease flares/complications in high-risk patients allocated to the Proactive arm versus the high-risk patients allocated to standard treatment

SECONDARY OUTCOMES:
Rate of disease flares/complications in low-risk patients | 24 months
  The rate of disease flares/complications in low-risk patients continuing their treatment unaltered compared to the high-risk patients allocated to the standard treatment arm.
Rate of mucosal healing | 24 months
  The rate of mucosal healing, defined as LS<350 for worst segment and LS<450 for total small bowel in the two high risk arms at 24 months
Rate of disease flares/complications compared to a previous similar study | 24 months
  The rate of disease flares/complications in low-risk and high-risk patients continuing their treatment unaltered compared to the rate in the patients enrolled in Sheba-IIRN previously completed study.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Eliakim, Prof., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba_Medical_Center, Tel Litwinsky, Israel

REFERENCES:
- [Derived] Margalit Yehuda R, Davidov Y, Selinger L, Ungar B, Lahat A, Yablecovitch D, Neuman S, Kopylov U, Ben Horin S, Eliakim R; Israeli IBD Research Nucleus (IIRN). The Visibility and Performance of Small Bowel Video Capsule Endoscopy With and Without Pre-Procedural Purge Preparation in the Same Patients. J Gastroenterol Hepatol. 2025 Jun;40(6):1485-1491. doi: 10.1111/jgh.16954. Epub 2025 Apr 3. PMID 40176636
- [Derived] Ben-Horin S, Lahat A, Ungar B, Ukashi O, Yablecovitch D, Amitai MM, Haberman Y, Selinger L, Talan-Asher A, Kriger-Sharabi O, Naftali T, Ron Y, Yanai H, Dotan I, Kopylov U, Eliakim R; Israeli IBD Research Nucleus (IIRN). Capsule Endoscopy-Guided Proactive Treat-to-Target Versus Continued Standard Care in Patients With Quiescent Crohn's Disease: A Randomized Controlled Trial. Gastroenterology. 2025 Jul;169(1):85-93.e3. doi: 10.1053/j.gastro.2025.02.031. Epub 2025 Mar 17. PMID 40107519